CLINICAL TRIAL: NCT02076919
Title: A Randomized, Double-Masked, Vehicle-Controlled, First-in-Human Study to Assess the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of Topically Delivered LHA510 in Elderly Subjects and Patients With Age-Related Macular Degeneration
Brief Title: First-in-Human Study of LHA510 in Elderly Subjects and Patients With Age-Related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: C-13-007
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Results first posted 2015-09-04 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Age-Related Macular Degeneration
Keywords: LHA510; First in human; Safety; Tolerability; Pharmacokinetics; Elderly; Age-Related Macular Degeneration; AMD; Ocular; Eye drop
MeSH Terms: conditions — Macular Degeneration | interventions — acrizanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- LHA510 Part 1 (Experimental): LHA510 Ophthalmic Suspension in 1 of 4 concentrations, 1 drop instilled in the study eye as a single dose during Part 1
  Interventions: Drug: LHA510 Ophthalmic Suspension
- LHA510 Vehicle Part 1 (Placebo Comparator): Inactive ingredients, 1 drop instilled in the study eye as a single dose during Part 1
  Interventions: Drug: LHA510 Vehicle
- LHA510 Part 2 (Experimental): LHA510 Ophthalmic Suspension in 1 of 4 concentrations, 1 drop instilled in the study eye once, twice, or three times daily for 7 days during Part 2
  Interventions: Drug: LHA510 Ophthalmic Suspension
- LHA510 Vehicle Part 2 (Placebo Comparator): Inactive ingredients, 1 drop instilled in the study eye once, twice, or 3 times daily for 7 days during Part 2
  Interventions: Drug: LHA510 Vehicle

INTERVENTIONS:
Drug: LHA510 Ophthalmic Suspension — Ophthalmic suspension in 4 concentration levels topically administered in Part 1 and Part 2
  Arms: LHA510 Part 1; LHA510 Part 2
Drug: LHA510 Vehicle — Inactive ingredients used for masking purposes
  Arms: LHA510 Vehicle Part 1; LHA510 Vehicle Part 2

SUMMARY:
The purpose of this first-in-human study is to assess the local ocular and systemic safety and tolerability of LHA510 eye drops when administered at various concentrations and dosing frequencies.

DETAILED DESCRIPTION:
This first-in-human study was conducted in two parts. Part 1 was a single ascending dose (SAD) design to assess the local ocular and systemic safety and tolerability of a single topical eye drop of LHA510 administered at various concentrations. Four separate cohorts of unique elderly subjects (55 to 80 years) were utilized, with each cohort randomized to receive either topical LHA510 or vehicle in a 3:1 ratio as a single dose. A disposition evaluation was performed 7 days later. Part 2 was a multiple ascending dose (MAD) design to assess the local ocular and systemic safety and tolerability of LHA510 administered at various concentrations and dosing frequencies. Six separate cohorts of unique AMD subjects were utilized, with each cohort randomized to receive either topical LHA510 or vehicle in a 3:1 ratio for 7 days. A disposition evaluation was performed 14 days after the first dose of study drug. A review of all available safety data was conducted by the Sponsor and the PI(s) prior to dose escalation (cohort progression). The same concentrations levels were used in Part 1 and Part 2 and are ordered as Lowest, Next Lowest, Next Highest, and Highest.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Vital signs within the following ranges:

  * oral body temperature between 35.0-37.5 °C
  * systolic blood pressure, 90-150 mm Hg
  * diastolic blood pressure, 50-90 mm Hg
  * pulse rate, 40 - 100 bpm.
* Weigh at least 50 kg.
* Able to communicate well with the investigator.
* Able to understand and comply with the requirements of the study.

Additional eligibility criteria for Part 2 (AMD subjects):

* Evidence of AMD in one or both eyes.
* Age 55-90.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any currently active ocular condition that requires use of topical eye drops.
* Use of contact lens over the course of the study.
* Abnormal corneal examination results at screening or eligibility.
* History of any ocular surgery within the past 6 months prior to study participation.
* Use of other investigational drugs within 30 days of enrollment.
* History of hypersensitivity or allergy to any of the study drugs (including fluorescein) or to drugs of similar chemical classes.
* History of clinically significant ECG abnormalities, or any ECG abnormality at screening or eligibility.
* Known history or current clinically significant arrhythmias.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential.
* Use of any prohibited medication as specified in the protocol.
* Donation or loss of 400 ml or more of blood within eight (8) weeks prior to initial dosing.
* Low hemoglobin levels at screening or eligibility as specified in the protocol.
* Significant illness as specified in the protocol.
* History of drug or alcohol abuse within the 12 months prior to dosing.

Additional exclusion criteria for Part 1 (healthy subjects):

* Abnormal thickness of the central retinal subfield on OCT at screening.
* History of any chronic eye disease other than refractive error, incipient cataract, strabismic amblyopia, or anisometropic amblyopia.

Additional exclusion criteria for Part 2 (AMD subjects):

* Any of the following treatments to the study eye within 28 days prior to dosing: ranibizumab (Lucentis®), aflibercept (Eylea®), bevacizumab (Avastin®), pegaptanib (Macugen®), or any other VEGF inhibitor.
* Patients who have required and received regular monthly injections of these drugs in the months preceding the study.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Maietta, BSc, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from a single investigational site located in the US.
Pre-assignment Details: Of the 110 enrolled, 30 subjects were exited as screen failures prior to randomization. This reporting group includes all randomized subjects (80).
Groups:
- LHA510, Part 1: Ophthalmic suspension in 1 of 4 concentrations, 1 drop instilled in the study eye as a single dose during Part 1
- Vehicle, Part 1: Inactive ingredients, 1 drop instilled in the study eye as a single dose during Part 1
- LHA510, Part 2: Ophthalmic suspension in 1 of 4 concentrations, 1 drop instilled in the study eye once, twice, or three times daily for 7 days during Part 2
- Vehicle, Part 2: Inactive ingredients, 1 drop instilled in the study eye once, twice, or 3 times daily for 7 days during Part 2
Period: Overall Study
Arm/Group | LHA510, Part 1 | Vehicle, Part 1 | LHA510, Part 2 | Vehicle, Part 2
Started | 24 | 8 | 36 | 12
Completed | 24 | 8 | 36 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all enrolled subjects.
Groups:
- LHA510 Lowest, Part 1; LHA510 Next Lowest, Part 1; LHA510 Next Highest, Part 1; LHA510 Highest, Part 1; Vehicle, Part 1: 1 drop instilled in the study eye as a single dose
- LHA510 Lowest, Part 2; LHA510 Next Lowest, Part 2; LHA510 Next Highest, Part 2; LHA510 Highest, Part 2: 1 drop instilled in the study eye once daily for 7 days
- LHA510 Highest BID, Part 2: 1 drop instilled in the study eye twice daily for 7 days
- LHA510 Highest TID, Part 2: 1 drop instilled in the study eye three times daily for 7 days
- Vehicle, Part 2: 1 drop instilled in the study eye once, twice, or three times daily for 7 days
- Total: Total of all reporting groups
Arm/Group | LHA510 Lowest, Part 1 | LHA510 Next Lowest, Part 1 | LHA510 Next Highest, Part 1 | LHA510 Highest, Part 1 | Vehicle, Part 1 | LHA510 Lowest, Part 2 | LHA510 Next Lowest, Part 2 | LHA510 Next Highest, Part 2 | LHA510 Highest, Part 2 | LHA510 Highest BID, Part 2 | LHA510 Highest TID, Part 2 | Vehicle, Part 2 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 80
Age, Customized [Number; unit: participants]
  55-64 years | 2 | 3 | 4 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 14
  ≥ 65 years | 4 | 3 | 2 | 4 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 12 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 4 | 4 | 4 | 3 | 2 | 3 | 3 | 2 | 8 | 41
  Male | 3 | 4 | 3 | 2 | 4 | 2 | 3 | 4 | 3 | 3 | 4 | 4 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Serious Adverse Event That, in the Opinion of the Investigator, is Related to the Study Drug, Part 1
Description: A serious adverse event (SAE) was defined as any event which is fatal or life-threatening, which requires or prolongs hospitalization, which is significantly or permanently disabling or incapacitating, which constitutes a congenital anomaly or a birth defect, or which is medically significant, may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: From time of consent until 30 days after stopping the trial/study drug
Population: This analysis population includes all enrolled subjects in Part 1.
Measure: Number; unit: participants
Arm/Group | LHA510 Lowest, Part 1 | LHA510 Next Lowest, Part 1 | LHA510 Next Highest, Part 1 | LHA510 Highest, Part 1 | Vehicle, Part 1
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Subjects With a Serious Adverse Event That, in the Opinion of the Investigator, is Related to the Study Drug, Part 2
Description: as for outcome 1
Time Frame: From time of consent until 30 days after stopping the trial/study drug
Population: This analysis population includes all enrolled subjects in Part 2.
Measure: Number; unit: participants
Arm/Group | LHA510 Lowest, Part 2 | LHA510 Next Lowest, Part 2 | LHA510 Next Highest, Part 2 | LHA510 Highest, Part 2 | LHA510 Highest BID, Part 2 | LHA510 Highest TID, Part 2 | Vehicle, Part 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: The Observed Maximum Plasma (or Serum or Blood) Concentration Following Drug Administration [Mass / Volume] (Cmax), Part 2
Description: Plasma concentrations were quantitated using a high performance liquid chromatography/tandem mass spectometry method.Timepoints of assessment for Arms 1-4 were Days 1 and 7: 0h (pre-dose), 0.25h, 0.5h, 1h, 2h, 4h, 6h, 8h, 12h and 24h post-dose; and Day 15: 0h. Timepoints of assessment for LHA Highest BID were Days 1 and 7: 0h (pre-dose), 0.25h, 0.5h, 1h, 2h, 4h, 6h, 8h and 12h post-dose; and Day 15: 0h. Timepoints of assessment for LHA510 Highest TID were Days 1 and 7: 0h (pre-dose), 0.25h, 0.5h, 1h, 2h, 4h, 0h (pre-2nd dose), 0.5h, 2h, 0h (pre-3rd dose), 0.25h, 0.5h, 1h, 2h, 4h, 12h post-dose; and Day 15: 0h.
Time Frame: Up to Day 15
Population: This analysis population includes all enrolled subjects in Part 2.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LHA510 Lowest, Part 2 | LHA510 Next Lowest, Part 2 | LHA510 Next Highest, Part 2 | LHA510 Highest, Part 2 | LHA510 Highest BID, Part 2 | LHA510 Highest TID, Part 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation.

4. Secondary Outcome: The Time to Reach the Maximum Concentration After Drug Administration [Time] (Tmax), Part 2
Description: Plasma concentrations were quantitated using a high performance liquid chromatography/tandem mass spectometry method. Timepoints of assessment for Arms 1-4 were Days 1 and 7: 0h (pre-dose), 0.25h, 0.5h, 1h, 2h, 4h, 6h, 8h, 12h and 24h post-dose; and Day 15: 0h. Timepoints of assessment for LHA Highest BID were Days 1 and 7: 0h (pre-dose), 0.25h, 0.5h, 1h, 2h, 4h, 6h, 8h and 12h post-dose; and Day 15: 0h. Timepoints of assessment for LHA510 Highest TID were Days 1 and 7: 0h (pre-dose), 0.25h, 0.5h, 1h, 2h, 4h, 0h (pre-2nd dose), 0.5h, 2h, 0h (pre-3rd dose), 0.25h, 0.5h, 1h, 2h, 4h, 12h post-dose; and Day 15: 0h.
Time Frame: Up to Day 15
Population: This analysis population includes all enrolled subjects in Part 2.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | LHA510 Lowest, Part 2 | LHA510 Next Lowest, Part 2 | LHA510 Next Highest, Part 2 | LHA510 Highest, Part 2 | LHA510 Highest BID, Part 2 | LHA510 Highest TID, Part 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hour | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation.

5. Secondary Outcome: The Area Under the Plasma (or Serum or Blood) Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration [Mass x Time/Volume] (AUClast), Part 2
Description: as for outcome 4
Time Frame: Up to Day 15
Population: This analysis population includes all enrolled subjects in Part 2.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | LHA510 Lowest, Part 2 | LHA510 Next Lowest, Part 2 | LHA510 Next Highest, Part 2 | LHA510 Highest, Part 2 | LHA510 Highest BID, Part 2 | LHA510 Highest TID, Part 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng*h/mL | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation.

6. Secondary Outcome: The Terminal Elimination Half-life [Time] (T1/2), Part 2
Description: as for outcome 4
Time Frame: Up to Day 15
Population: This analysis population includes all enrolled subjects in Part 2.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | LHA510 Lowest, Part 2 | LHA510 Next Lowest, Part 2 | LHA510 Next Highest, Part 2 | LHA510 Highest, Part 2 | LHA510 Highest BID, Part 2 | LHA510 Highest TID, Part 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hour | NA (NA) — The analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — The analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — The analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — The analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — The analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — The analysis was not conducted because the concentration was too low to allow reliable estimation.

7. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Each Post Dose Timepoint, Part 1
Description: Diastolic blood pressure (pressure in the arteries when the heart rests between beats) was measured using an automated validated device, with an appropriately sized cuff, and assessed in the sitting position after the subject had rested for at least 3 minutes, and again (when required) after 3 minutes in the standing position.
Time Frame: Day 1: 0.25h, 0.5h, 1h, 2h, 4h, 6h, 8h, 12h and 24h post-dose
Population: This analysis population includes all enrolled subjects in Part 1.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LHA510 Lowest, Part 1 | LHA510 Next Lowest, Part 1 | LHA510 Next Highest, Part 1 | LHA510 Highest, Part 1 | Vehicle, Part 1
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
mmHg
  Day 1, 0.25 hours | 5.2 (3.19) | -5.5 (3.35) | 2.8 (3.14) | 4.1 (3.12) | -5.2 (2.70)
  Day 1, 0.50 hours | 3.4 (3.19) | -0.2 (3.35) | 5.6 (3.14) | 7.6 (3.12) | 2.1 (2.70)
  Day 1, 1.00 hours | 3.9 (3.19) | 2.2 (3.35) | 5.3 (3.14) | 5.1 (3.12) | -1.4 (2.70)
  Day 1, 2.00 hours | -3.8 (3.19) | -1.0 (3.35) | -1.6 (3.14) | -0.9 (3.12) | -6.5 (2.70)
  Day 1, 4.00 hours | 5.4 (3.19) | 3.7 (3.35) | 4.3 (3.14) | 4.1 (3.12) | 2.4 (2.70)
  Day 1, 6.00 hours | -1.1 (3.19) | 1.2 (3.35) | 2.9 (3.14) | 3.1 (3.12) | -6.1 (2.70)
  Day 1, 8.00 hours | 3.6 (3.19) | 1.5 (3.35) | 4.6 (3.14) | 2.5 (3.12) | 0.0 (2.70)
  Day 1, 12.00 hours | 3.7 (3.19) | 1.7 (3.35) | 4.1 (3.14) | -2.2 (3.12) | -3.9 (2.70)
  Day 1, 24.00 hours | 8.2 (3.19) | 5.5 (3.35) | 6.1 (3.14) | 5.3 (3.12) | 4.0 (2.70)

8. Primary Outcome: Number of Subjects Experiencing a Non-serious Adverse Event, Part I
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. An AE, therefore, could be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the study treatment, whether or not related to the treatment.
Time Frame: From time of consent until 30 days after stopping the trial/study drug
Population: This analysis population includes all enrolled subjects in Part 1.
Measure: Number; unit: participants
Arm/Group | LHA510 Lowest, Part 1 | LHA510 Next Lowest, Part 1 | LHA510 Next Highest, Part 1 | LHA510 Highest, Part 1 | Vehicle, Part 1
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants | 2 | 1 | 0 | 1 | 1

9. Primary Outcome: Number of Subjects Experiencing a Non-serious Adverse Event, Part 2
Description: as for outcome 8
Time Frame: From time of consent until 30 days after stopping the trial/study drug
Population: This analysis population includes all enrolled subjects in Part 2.
Measure: Number; unit: participants
Arm/Group | LHA510 Lowest, Part 2 | LHA510 Next Lowest, Part 2 | LHA510 Next Highest, Part 2 | LHA510 Highest, Part 2 | LHA510 Highest BID, Part 2 | LHA510 Highest TID, Part 2 | Vehicle, Part 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
participants | 3 | 1 | 1 | 2 | 2 | 1 | 3

10. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Each Post Dose Timepoint, Part 1
Description: Systolic blood pressure (pressure when the heart is contracting) was measured using an automated validated device, with an appropriately sized cuff, and assessed in the sitting position after the subject had rested for at least 3 minutes, and again (when required) after 3 minutes in the standing position.
Time Frame: Day 1: 0.25h, 0.5h, 1h, 2h, 4h, 6h, 8h, 12h and 24h post-dose
Population: This analysis population includes all enrolled subjects in Part 1.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LHA510 Lowest, Part 1 | LHA510 Next Lowest, Part 1 | LHA510 Next Highest, Part 1 | LHA510 Highest, Part 1 | Vehicle, Part 1
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
mmHg
  Day 1, 0.25 hours | 4.7 (5.00) | 0.5 (5.11) | 0.5 (5.05) | 5.3 (4.97) | 0.2 (4.32)
  Day 1, 0.50 hours | -1.3 (5.00) | 0.1 (5.11) | -0.3 (5.05) | 6.9 (4.97) | 4.9 (4.32)
  Day 1, 1.00 hours | 1.7 (5.00) | 2.8 (5.11) | 1.2 (5.05) | 2.9 (4.97) | 4.4 (4.32)
  Day 1, 2.00 hours | -4.6 (5.00) | 5.3 (5.11) | 0.5 (5.05) | 9.8 (4.97) | 1.3 (4.32)
  Day 1, 4.00 hours | -6.3 (5.00) | 9.3 (5.11) | 4.7 (5.05) | 5.4 (4.97) | -0.9 (4.32)
  Day 1, 6.00 hours | -2.0 (5.00) | 10.5 (5.11) | 0.7 (5.05) | 4.9 (4.97) | -4.6 (4.32)
  Day 1, 8.00 hours | 4.0 (5.00) | 4.3 (5.11) | 2.2 (5.05) | 14.1 (4.97) | -2.6 (4.32)
  Day 1, 12.00 hours | 3.9 (5.00) | 11.8 (5.11) | -3.0 (5.05) | 5.3 (4.97) | -1.9 (4.32)
  Day 1, 24.00 hours | 9.4 (5.00) | 9.6 (5.11) | 2.3 (5.05) | 8.9 (4.97) | 2.1 (4.32)

11. Secondary Outcome: Change From Baseline in Mean Arterial Blood Pressure at Each Post Dose Timepoint, Part 1
Description: Mean arterial blood pressure (average pressure in the arteries during one cardiac cycle) was measured using an automated validated device, with an appropriately sized cuff, and assessed in the sitting position after the subject had rested for at least 3 minutes, and again (when required) after 3 minutes in the standing position.
Time Frame: Day 1: 0.25h, 0.5h, 1h, 2h, 4h, 6h, 8h, 12h and 24h post-dose
Population: This analysis population includes all enrolled subjects in Part 1.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LHA510 Lowest, Part 1 | LHA510 Next Lowest, Part 1 | LHA510 Next Highest, Part 1 | LHA510 Highest, Part 1 | Vehicle, Part 1
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
mmHg
  Day 1, 0.25 hours | 5.2 (3.25) | -4.4 (3.52) | 2.4 (3.31) | 4.7 (3.26) | -3.4 (2.81)
  Day 1, 0.50 hours | 2.0 (3.25) | -0.9 (3.52) | 4.0 (3.31) | 7.6 (3.26) | 3.1 (2.81)
  Day 1, 1.00 hours | 3.3 (3.25) | 1.5 (3.52) | 4.3 (3.31) | 4.6 (3.26) | 0.6 (2.81)
  Day 1, 2.00 hours | -3.9 (3.25) | 0.3 (3.52) | -0.5 (3.31) | 2.9 (3.26) | -3.9 (2.81)
  Day 1, 4.00 hours | 1.7 (3.25) | 4.7 (3.52) | 4.8 (3.31) | 4.8 (3.26) | 1.3 (2.81)
  Day 1, 6.00 hours | -1.2 (3.25) | 3.4 (3.52) | 2.6 (3.31) | 4.0 (3.26) | -5.6 (2.81)
  Day 1, 8.00 hours | 3.9 (3.25) | 1.6 (3.52) | 4.2 (3.31) | 6.6 (3.26) | -0.8 (2.81)
  Day 1, 12.00 hours | 3.9 (3.25) | 4.2 (3.52) | 2.2 (3.31) | 0.5 (3.26) | -3.2 (2.81)
  Day 1, 24.00 hours | 8.8 (3.25) | 6.0 (3.52) | 5.3 (3.31) | 6.7 (3.26) | 3.4 (2.81)

12. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Each Post Dose Timepoint, Part 2
Description: as for outcome 7
Time Frame: Day 1 and 7: 0.25h, 0.5h, 1h, 2h, 4h, 6h, 8h, 12h and 24h post-dose
Population: This analysis population includes all enrolled subjects in Part 2.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LHA510 Lowest, Part 2 | LHA510 Next Lowest, Part 2 | LHA510 Next Highest, Part 2 | LHA510 Highest, Part 2 | LHA510 Highest BID, Part 2 | LHA510 Highest TID, Part 2 | Vehicle, Part 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
mmHg
  Day 1, 0.25 Hours | -1.0 (2.94) | -4.4 (2.96) | -0.6 (2.95) | -2.9 (2.93) | 2.5 (2.93) | 0.6 (2.93) | -0.5 (2.07)
  Day 1, 0.50 Hours | -1.7 (2.94) | -7.2 (2.96) | -4.5 (2.95) | -4.6 (2.93) | 4.3 (2.93) | -2.2 (2.93) | 2.4 (2.07)
  Day 1, 1.00 Hours | 4.3 (2.94) | -7.7 (2.96) | 0.2 (2.95) | 1.9 (2.93) | 1.7 (2.93) | -5.4 (2.93) | 0.3 (2.07)
  Day 1, 2.00 Hours | -9.4 (2.94) | -6.5 (2.96) | 1.2 (2.95) | -4.1 (2.93) | -4.2 (2.93) | -6.7 (2.93) | -4.9 (2.07)
  Day 1, 4.00 Hours | 1.8 (2.94) | -4.0 (2.96) | -5.5 (2.95) | 0.9 (2.93) | -1.2 (2.93) | -2.4 (2.93) | -0.2 (2.07)
  Day 1, 6.00 Hours | -4.9 (2.94) | -6.9 (2.96) | -3.3 (2.95) | -4.1 (2.93) | -2.2 (2.93) | -5.9 (2.93) | -5.3 (2.07)
  Day 1, 8.00 Hours | 3.1 (2.94) | 2.1 (2.96) | -2.0 (2.95) | 1.4 (2.93) | 4.3 (2.93) | 1.3 (2.93) | 5.7 (2.07)
  Day 1, 12.00 Hours | 2.3 (2.94) | 1.0 (2.96) | -1.3 (2.95) | -2.1 (2.93) | 7.2 (2.93) | -0.4 (2.93) | 0.4 (2.07)
  Day 1, 24.00 Hours | 3.8 (2.94) | -2.5 (2.96) | 3.9 (2.95) | 2.3 (2.93) | -2.7 (2.93) | -0.7 (2.93) | 2.7 (2.07)
  Day 7, 0.25 Hours | -3.4 (2.94) | -6.2 (2.96) | -3.3 (2.95) | -1.7 (2.93) | -2.8 (2.93) | -2.4 (2.93) | -3.6 (2.07)
  Day 7, 0.50 Hours | -5.9 (2.94) | -5.7 (2.96) | -10.0 (2.95) | -2.1 (2.93) | -3.2 (2.93) | 1.6 (2.93) | -2.8 (2.07)
  Day 7, 1.00 Hours | -6.0 (2.94) | -4.9 (2.96) | -4.3 (2.95) | -3.1 (2.93) | -6.5 (2.93) | -2.2 (2.93) | -2.9 (2.07)
  Day 7, 2.00 Hours | -4.2 (2.94) | -6.4 (2.96) | -8.3 (2.95) | -4.7 (2.93) | -0.7 (2.93) | -5.4 (2.93) | -9.6 (2.07)
  Day 7, 4.00 Hours | -6.0 (2.94) | -6.7 (2.96) | -9.3 (2.95) | -3.6 (2.93) | -8.2 (2.93) | -2.4 (2.93) | -7.8 (2.07)
  Day 7, 6.00 Hours | -4.4 (2.94) | 0.3 (2.96) | -10.3 (2.95) | -5.6 (2.93) | -8.8 (2.93) | -6.4 (2.93) | -5.3 (2.07)
  Day 7, 8.00 Hours | -0.7 (2.94) | 1.0 (2.96) | -6.1 (2.95) | -2.7 (2.93) | -3.0 (2.93) | 1.3 (2.93) | -2.4 (2.07)
  Day 7, 12.00 Hours | -9.5 (2.94) | -1.0 (2.96) | -7.1 (2.95) | -3.7 (2.93) | -2.3 (2.93) | -2.7 (2.93) | -3.0 (2.07)
  Day 7, 24.00 Hours | -4.2 (2.94) | -2.2 (2.96) | -7.5 (2.95) | -3.7 (2.93) | -1.2 (2.93) | -1.4 (2.93) | 0.4 (2.07)

13. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Each Post Dose Timepoint, Part 2
Description: as for outcome 10
Time Frame: Day 1 and 7: 0.25h, 0.5h, 1h, 2h, 4h, 6h, 8h, 12h and 24h post-dose
Population: This analysis population includes all enrolled subjects in Part 2.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LHA510 Lowest, Part 2 | LHA510 Next Lowest, Part 2 | LHA510 Next Highest, Part 2 | LHA510 Highest, Part 2 | LHA510 Highest BID, Part 2 | LHA510 Highest TID, Part 2 | Vehicle, Part 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
mmHg
  Day 1, 0.25 Hours | 12.5 (5.70) | -11.1 (5.90) | -4.1 (5.70) | -4.8 (5.74) | 0.6 (5.72) | -4.1 (5.69) | 1.0 (4.03)
  Day 1, 0.50 Hours | -3.9 (5.70) | -12.7 (5.90) | -0.4 (5.70) | -11.4 (5.74) | -5.4 (5.72) | -5.8 (5.69) | 0.8 (4.03)
  Day 1, 1.00 Hours | 7.1 (5.70) | -13.1 (5.90) | 3.4 (5.70) | -8.9 (5.74) | -3.1 (5.72) | -8.9 (5.69) | 0.8 (4.03)
  Day 1, 2.00 Hours | -0.7 (5.70) | -3.9 (5.90) | -0.9 (5.70) | -6.4 (5.74) | -5.6 (5.72) | -10.6 (5.69) | -4.6 (4.03)
  Day 1, 4.00 Hours | 5.3 (5.70) | -5.4 (5.90) | -9.9 (5.70) | 0.7 (5.74) | -3.4 (5.72) | -0.4 (5.69) | -0.4 (4.03)
  Day 1, 6.00 Hours | -3.2 (5.70) | -15.6 (5.90) | -8.6 (5.70) | 0.4 (5.74) | -2.2 (5.72) | -6.9 (5.69) | -10.1 (4.03)
  Day 1, 8.00 Hours | 5.5 (5.70) | 11.1 (5.90) | -9.8 (5.70) | -1.4 (5.74) | -6.1 (5.72) | 6.1 (5.69) | 5.1 (4.03)
  Day 1, 12.00 Hours | 5.5 (5.70) | 11.8 (5.90) | -8.8 (5.70) | -3.9 (5.74) | 3.4 (5.72) | 1.2 (5.69) | 5.9 (4.03)
  Day 1, 24.00 Hours | 5.0 (5.70) | 0.1 (5.90) | -2.6 (5.70) | 7.7 (5.74) | -6.9 (5.72) | -6.8 (5.69) | 2.6 (4.03)
  Day 7, 0.25 Hours | -5.0 (5.70) | -7.6 (5.90) | -9.4 (5.70) | -2.3 (5.74) | -13.7 (5.72) | -11.3 (5.69) | -3.3 (4.03)
  Day 7, 0.50 Hours | -5.7 (5.70) | -6.2 (5.90) | -14.9 (5.70) | -8.8 (5.74) | -9.9 (5.72) | -9.9 (5.69) | -6.4 (4.03)
  Day 7, 1.00 Hours | -1.2 (5.70) | -9.4 (5.90) | -9.4 (5.70) | -4.6 (5.74) | -18.6 (5.72) | -6.1 (5.69) | -3.9 (4.03)
  Day 7, 2.00 Hours | -5.4 (5.70) | -6.9 (5.90) | -9.8 (5.70) | -6.1 (5.74) | -14.7 (5.72) | -0.4 (5.69) | -12.3 (4.03)
  Day 7, 4.00 Hours | -4.2 (5.70) | -5.1 (5.90) | -12.4 (5.70) | -3.8 (5.74) | -9.4 (5.72) | -8.9 (5.69) | -17.4 (4.03)
  Day 7, 6.00 Hours | -0.4 (5.70) | 4.3 (5.90) | -18.8 (5.70) | -6.6 (5.74) | -7.7 (5.72) | -5.4 (5.69) | -3.3 (4.03)
  Day 7, 8.00 Hours | 0.1 (5.70) | 15.6 (5.90) | -9.8 (5.70) | 0.6 (5.74) | -10.9 (5.72) | 0.1 (5.69) | -0.9 (4.03)
  Day 7, 12.00 Hours | -4.5 (5.70) | 8.4 (5.90) | -10.9 (5.70) | -9.6 (5.74) | -7.6 (5.72) | -4.9 (5.69) | -5.5 (4.03)
  Day 7, 24.00 Hours | -0.5 (5.70) | 0.6 (5.90) | -23.1 (5.70) | -4.4 (5.74) | -4.4 (5.72) | 0.6 (5.69) | 7.3 (4.03)

14. Secondary Outcome: Change From Mean Arterial Blood Pressure at Each Post Dose Timepoint, Part 2
Description: as for outcome 11
Time Frame: Day 1 and 7: 0.25h, 0.5h, 1h, 2h, 4h, 6h, 8h, 12h and 24h post-dose
Population: This analysis population includes all enrolled subjects in Part 2.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Groups:
- Vehicle, Part 2: One drop instilled in the study eye once, twice, or three times daily for 7 days
Arm/Group | LHA510 Lowest, Part 2 | LHA510 Next Lowest, Part 2 | LHA510 Next Highest, Part 2 | LHA510 Highest, Part 2 | LHA510 Highest BID, Part 2 | LHA510 Highest TID, Part 2 | Vehicle, Part 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
mmHg
  Day 1, 0.25 Hours | 3.5 (3.34) | -6.8 (3.41) | -1.7 (3.35) | -3.5 (3.33) | 1.9 (3.33) | -1.0 (3.33) | -0.0 (2.35)
  Day 1, 0.50 Hours | -2.4 (3.34) | -9.2 (3.41) | -3.1 (3.35) | -6.8 (3.33) | 1.1 (3.33) | -3.4 (3.33) | 1.8 (2.35)
  Day 1, 1.00 Hours | 5.3 (3.34) | -9.7 (3.41) | 1.3 (3.35) | -1.6 (3.33) | 0.1 (3.33) | -6.6 (3.33) | 0.4 (2.35)
  Day 1, 2.00 Hours | -6.4 (3.34) | -5.8 (3.41) | 0.6 (3.35) | -4.8 (3.33) | -4.6 (3.33) | -8.1 (3.33) | -4.8 (2.35)
  Day 1, 4.00 Hours | 3.0 (3.34) | -4.7 (3.41) | -6.9 (3.35) | 0.9 (3.33) | -1.9 (3.33) | -1.8 (3.33) | -0.3 (2.35)
  Day 1, 6.00 Hours | -4.3 (3.34) | -10.0 (3.41) | -5.0 (3.35) | -2.5 (3.33) | -2.1 (3.33) | -6.3 (3.33) | -6.9 (2.35)
  Day 1, 8.00 Hours | 4.0 (3.34) | 4.9 (3.41) | -4.5 (3.35) | 0.5 (3.33) | 0.9 (3.33) | 2.8 (3.33) | 5.5 (2.35)
  Day 1, 12.00 Hours | 3.4 (3.34) | 4.4 (3.41) | -3.7 (3.35) | -2.6 (3.33) | 6.0 (3.33) | 0.1 (3.33) | 2.2 (2.35)
  Day 1, 24.00 Hours | 4.2 (3.34) | -1.8 (3.41) | 1.8 (3.35) | 4.1 (3.33) | -4.0 (3.33) | -2.8 (3.33) | 2.6 (2.35)
  Day 7, 0.25 Hours | -3.9 (3.34) | -6.8 (3.41) | -5.3 (3.35) | -1.9 (3.33) | -6.4 (3.33) | -5.4 (3.33) | -3.5 (2.35)
  Day 7, 0.50 Hours | -5.8 (3.34) | -6.1 (3.41) | -11.6 (3.35) | -4.3 (3.33) | -5.4 (3.33) | -2.3 (3.33) | -4.0 (2.35)
  Day 7, 1.00 Hours | -4.4 (3.34) | -6.6 (3.41) | -5.9 (3.35) | -3.5 (3.33) | -10.5 (3.33) | -3.6 (3.33) | -3.3 (2.35)
  Day 7, 2.00 Hours | -4.5 (3.34) | -6.7 (3.41) | -8.7 (3.35) | -5.1 (3.33) | -5.3 (3.33) | -3.8 (3.33) | -10.5 (2.35)
  Day 7, 4.00 Hours | -5.4 (3.34) | -6.3 (3.41) | -10.3 (3.35) | -3.6 (3.33) | -8.5 (3.33) | -4.6 (3.33) | -11.0 (2.35)
  Day 7, 6.00 Hours | -3.0 (3.34) | 1.4 (3.41) | -13.1 (3.35) | -5.9 (3.33) | -8.4 (3.33) | -6.1 (3.33) | -4.6 (2.35)
  Day 7, 8.00 Hours | -0.4 (3.34) | 5.7 (3.41) | -7.3 (3.35) | -1.6 (3.33) | -5.6 (3.33) | 0.8 (3.33) | -1.9 (2.35)
  Day 7, 12.00 Hours | -7.8 (3.34) | 1.9 (3.41) | -8.3 (3.35) | -5.6 (3.33) | -4.0 (3.33) | -3.5 (3.33) | -3.8 (2.35)
  Day 7, 24.00 Hours | -2.9 (3.34) | -1.5 (3.41) | -12.6 (3.35) | -3.9 (3.33) | -2.2 (3.33) | -0.8 (3.33) | 2.7 (2.35)

ADVERSE EVENTS:
Time Frame: AEs were collected for the duration of the study (Feb 2014 - Jun 2014). This analysis group includes all enrolled subjects.
Description: An AE is defined as any untoward medical occurrence in a patient who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. AEs were obtained as solicited comments from the study subjects and observations by the study Investigator, as outlined in the study protocol.
Arm/Group | LHA510 Lowest, Part 1 | LHA510 Next Lowest, Part 1 | LHA510 Next Highest, Part 1 | LHA510 Highest, Part 1 | Vehicle, Part 1 | LHA510 Lowest, Part 2 | LHA510 Next Lowest, Part 2 | LHA510 Next Highest, Part 2 | LHA510 Highest, Part 2 | LHA510 Highest BID, Part 2 | LHA510 Highest TID, Part 2 | Vehicle, Part 2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 2/6 | 1/6 | 0/6 | 1/6 | 1/8 | 3/6 | 1/6 | 1/6 | 2/6 | 2/6 | 1/6 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LHA510 Lowest, Part 1 (N=6) | LHA510 Next Lowest, Part 1 (N=6) | LHA510 Next Highest, Part 1 (N=6) | LHA510 Highest, Part 1 (N=6) | Vehicle, Part 1 (N=8) | LHA510 Lowest, Part 2 (N=6) | LHA510 Next Lowest, Part 2 (N=6) | LHA510 Next Highest, Part 2 (N=6) | LHA510 Highest, Part 2 (N=6) | LHA510 Highest BID, Part 2 (N=6) | LHA510 Highest TID, Part 2 (N=6) | Vehicle, Part 2 (N=12)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye Pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion Site Irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombophlebitis Superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry Eye (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel Puncture Site Swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.